CLINICAL TRIAL: NCT01204970
Title: Confocal Laser Micro-endoscopy: New Insights in COPD and Lung Transplant Recipients
Brief Title: Confocal Laser Micro-endoscopy in Chronic Obstructive Pulmonary Disease (COPD) and Lung Transplant Recipients
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Marc Decramer, Prof. Dr., KU Leuven
Other Study IDs: B32220109292
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Lung Transplantation; Chronic Obstructive Pulmonary Disease
Keywords: Confocal Laser Scanning Microendoscopy; Small airways; COPD; Lung transplantation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- COPD: COPD Gold class 1-4
- Transplant: Lung transplant recipients
- Control: Patients with normal spirometric data

SUMMARY:
Aspects of confocal laser micro-endoscopy (CLME) and morphometry in chronic obstructive pulmonary disease (COPD) and lung transplant recipients is described and will be correlated with clinical findings in order to described small airway remodelling in these patients.

DETAILED DESCRIPTION:
In early phases of COPD, changes in small airway characteristics may develop. Elastin decay and matrix remodelling could be responsible for these changes. Using CLME changes of in the bronchiolar wall and alveolar ducts can be visualized, described and measured.

In lung transplant recipients, CMLE will be performed to distinguish characteristics of distal airways in stabile patient in contrast to patients with bronchiolitis obliterans syndrome.

In both groups data will be correlated with CT findings, pulmonary function tests and anatomopathological results.

ELIGIBILITY:
Inclusion Criteria:

* referral for bronchoscopic investigation/sampling
* informed consent signed
* recent spirometric data

Exclusion Criteria:

* sedated and/or ventilated patients
* patients on ICU
* patients under oral anticoagulation
* co-existing lung disease
* acute infectious pulmonary disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for a bronchoscopic procedure will be asked to undergo CLME. 3 pools will be made: COPD patients according to their pulmonary function test, lung transplant recipients and patients with normal spirometric results. In all groups the difference between active smokers and no-smokers will be made.
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2010-09; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
morphometry | 90 - 180 - 360 - 540 - 720 days
  morpohometrical analysis at different time point after lung transplantation

SECONDARY OUTCOMES:
adverse events | 90 - 180 - 360- 540- 720 days
  bleeding, pneumothorax, pleuritic chest pain during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Yserbyt, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Chistophe Dooms, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Marc Decramer, MD, PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven; Geert Verleden, Md, PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven; Wim Janssens, MD, PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Yserbyt J, Dooms C, Janssens W, Verleden GM. Endoscopic advanced imaging of the respiratory tract: exploring probe-based confocal laser endomicroscopy in emphysema. Thorax. 2018 Feb;73(2):188-190. doi: 10.1136/thoraxjnl-2016-209746. Epub 2017 Apr 14. PMID 28411249